CLINICAL TRIAL: NCT02017808
Title: A Prospective, Observational, Single-blinded, Longitudinal Optical Coherence Tomography Study of Effect of Copaxone (Glatiramer Acetate) on Retinal Nerve Fiber Layer Thickness in Patients With Relapsing-remitting Multiple Sclerosis Over 24 Months
Brief Title: Studying the Effects of Copaxone on Retinal Health Using Optical Tomography Over 24 Months
Acronym: GAO
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: GA-OCT
Record Dates: First submitted 2013-12-04; First posted 2013-12-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
Keywords: OCT; Copaxone; Multiple sclerosis; relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Copaxone: Patients with multiple sclerosis who are currently prescribed glatiramer acitate (Copaxone)
- OCT: Healthy controls

SUMMARY:
This is a prospective, observational, single-blinded, longitudinal, 24-month OCT study of the evolution of axonal loss, as evidenced by loss of RNFLT and TMV, in RRMS patients treated with GA and in healthy controls.

DETAILED DESCRIPTION:
The primary aim of this study is to explore whether treatment with Copaxone may decrease accumulation of axonal loss, as measured by retinal nerve fiber layer thickness (RNFLT) on optical coherence tomography (OCT) in patients with RRMS over 24 months and compared to a reference population of healthy controls.

The secondary objective of this study is to investigate the effect of GA on total macular volume (TMV) on OCT in patients with RRMS over 24 months. We will also explore how the 24-month changes of RNFLT and TMV on OCT relate to progression of disability, as measured by Expanded Disability Status Scale (EDSS).

ELIGIBILITY:
Inclusion Criteria:

* MS patients diagnosed with clinically definite MS according to the McDonald criteria (Polman et al., 2005)
* Starting GA monotherapy (20mg/day sc) at the time of the OCT scan
* Having baseline clinical OCT scan that included RNFLT and TMV assessment at the start of the GA
* Having baseline clinical OCT scan that included RNFLT and TMV assessment (healthy controls)
* MS patients having a RR disease course (Lublin and Reingold, 1996)
* Age 18-65 (healthy controls will be matched to MS patients for age and sex)
* Signed informed consent at the 24-month follow-up
* None of the exclusion criteria

Exclusion Criteria:

* Patients who had a relapse within 30 days prior to OCT scan date
* Patients who received steroid treatment within 30 days prior to OCT scan date
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study
* MS patients who used other imunomodulatory or immunosuppressant treatment other than GA during the follow-up (e.g., IFN-β, mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine, total body, azathioprine, methotrexate, IVIG, cellcept, natalizumab, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing remitting multiple sclerosis Healthy controls without known neurological problems.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Retinal health in multiple sclerosis patients prescribed copaxone | 24 months
  Participants will have an OCT retinal health will be determined by degree of axonal loss.

SECONDARY OUTCOMES:
Measuring disability progression | 24 months
  Investigating the effect of copaxone on total macular volume on OCT in patients with RRMS. Exploring progression of disability as measured by Expanded Disability Status Scale (EDSS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — SUNY University at Buffalo
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States